CLINICAL TRIAL: NCT02829593
Title: Measurement of Glucose Metabolism in Humans Using Magnetic Resonance at 7 Tesla: Effect of Recurrent Hypoglycemia on Hypothalamic GABA
Brief Title: Measurement of Glucose Metabolism in Humans: Effect of Recurrent Hypoglycemia on Hypothalamic GABA
Acronym: GABA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1511M80568
Record Dates: First submitted 2016-06-08; First posted 2016-07-12 (Estimated); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Type 1 Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- type 1 diabetes (Experimental): type 1 diabetes >5 years duration
  Interventions: Other: hypoglycemia (low blood sugar) and MRI
- healthy controls (Placebo Comparator)
  Interventions: Other: hypoglycemia (low blood sugar) and MRI

INTERVENTIONS:
Other: hypoglycemia (low blood sugar) and MRI — hypoglycemia (low blood sugar) and MRI

SUMMARY:
You are invited to participate in a study designed to investigate the effects of diabetes mellitus, high and low glucose, and high blood insulin on the brain. You were selected as a possible participant because you fit into one of the following categories. a) you are either healthy and competent, are not pregnant and you have no known medical disease and therefore your glucose metabolism will be typical of a normal person, or b) you have diabetes.

DETAILED DESCRIPTION:
Glucose is a major fuel for most organs in the human body, particularly the brain. How and where the body uses glucose is regulated by a number of hormones, for instance insulin and glucagon. In a number of diseases, in particular diabetes mellitus, the glucose supply to the brain may be different than normal, which may be a cause for reduced glucose awareness.

The purpose of this study is to determine the effects of altered glucose metabolism on the brain. For example, patients with long duration diabetes mellitus lose their ability to secrete the hormones necessary to protect them against hypoglycemia, which may be due to alterations in glucose availability to the human brain.

To measure these effects, we will use intravenous infusions of glucose and insulin.

ELIGIBILITY:
Inclusion Criteria:

* well controlled type 1 diabetes (hemoglobin A1c <7.5%)
* age 18-65
* healthy controls

Exclusion Criteria:

* history of stroke, seizures, neurosurgical procedures, or arrhythmias
* use of drugs that can alter GABA metabolism (such as benzodiazepines).
* Subjects must also meet requirements for a study in the magnet, which includes weight less than 300 lbs and the absence of metallic substances in their body.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Euglycemic GABA level in hypothalamus using MRI | Baseline to 2 month
  MRI measurement of GABA in the hypothalamus

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States